CLINICAL TRIAL: NCT05067478
Title: Composur, a Patient-centric, Phase IV, Open-label, Prospective, Real World US Study to Evaluate Vibegron on Patient Treatment Satisfaction, Quality of Life, and Healthcare Resource Utilization in Overactive Bladder
Brief Title: Composur: Study to Understand the Performance of Vibegron in Participants with Overactive Bladder (OAB)
Status: Completed | Type: Observational
Sponsor: Urovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: URO-901-4001
Record Dates: First submitted 2021-09-14; First posted 2021-10-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Overactive Bladder
Keywords: Vibegron; Urinary bladder, overactive; Beta-3 adrenergic receptor (β3-AR) agonists; Urge urinary incontinence; OAB
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Cohort A Vibegron: Participants with previous anticholinergic therapy experience will receive vibegron as per the United States (U.S.) label.
  Interventions: Drug: Vibegron
- Cohort B Vibegron: Participants with previous mirabegron monotherapy or mirabegron plus solifenacin or combination therapy experience will receive vibegron as per the U.S. label.
  Interventions: Drug: Vibegron

INTERVENTIONS:
Drug: Vibegron — Vibegron to be administered.
  Other Names: GEMTESA

SUMMARY:
This study will evaluate the treatment satisfaction, discontinuation, reasons for discontinuation, quality of life, healthcare resource utilization, and safety with Vibegron for the treatment of OAB in the context of real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of overactive bladder (OAB) with or without urgency urinary incontinence
* Symptoms of OAB for at least 3 months prior to the Baseline Visit
* Willing and able to complete electronic patient-reported outcomes questionnaires monthly for a minimum of 1 year
* Previous exposure to anticholinergics or mirabegron monotherapy and/or mirabegron plus solifenacin combination therapy prior to initiation of vibegron

Exclusion Criteria:

* Any contraindication to the use of vibegron per the United States label
* History of OAB treatment with botulinum toxin A; sacral neuromodulation; percutaneous tibial nerve stimulation; external beam radiation therapy; urinary stents within the last 6 months; pelvic or lower urinary tract surgery within the last 6 months; and urethral catheterizations within the last 3 months prior to the Baseline Visit
* History of mixed incontinence where stress incontinence is the predominant form (as determined by the investigator)
* Participants at risk of urinary retention (as determined by the investigator)
* Neurologic conditions associated with OAB symptoms, e.g., multiple sclerosis
* Pregnant or breastfeeding or plans to do so during the study
* Use of vibegron prior to the Baseline Visit either prescribed or in a previous vibegron clinical trial where the participant was on vibegron
* Anyone who, at the discretion of the investigator, is not suitable for treatment with a beta 3 agonist for OAB for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from primary care settings such as Family Practice, Urogynecology, and Urology practices
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Mean Satisfaction Domain Score as Assessed by the Overactive Bladder Satisfaction with Treatment Questionnaire (OAB-SAT-q) | Month 3
  The OAB-SAT-q is an 11-item questionnaire designed to assess participant's satisfaction with overactive bladder treatment in the clinical setting. It includes 3 subscales (satisfaction, side effects, endorsement) and 2 single-item assessments (convenience, preference), with a 4-week recall period. The OAB-SAT-q is scored by domains ranging from 0-100. Scores for the Convenience item range from 0-100. The Preference item is calculated as a percentage. Higher scores indicate higher levels of treatment satisfaction, endorsement, and convenience.
Mean Satisfaction Domain Score as Assessed by the OAB-SAT-q | Month 6
  The OAB-SAT-q is an 11-item questionnaire designed to assess participant's satisfaction with overactive bladder treatment in the clinical setting. It includes 3 subscales (satisfaction, side effects, endorsement) and 2 single-item assessments (convenience, preference), with a 4-week recall period. The OAB-SAT-q is scored by domains ranging from 0-100. Scores for the Convenience item range from 0-100. The Preference item is calculated as a percentage. Higher scores indicate higher levels of treatment satisfaction, endorsement, and convenience.
Mean Satisfaction Domain Score as Assessed by the OAB-SAT-q | Month 12
  The OAB-SAT-q is an 11-item questionnaire designed to assess participant's satisfaction with overactive bladder treatment in the clinical setting. It includes 3 subscales (satisfaction, side effects, endorsement) and 2 single-item assessments (convenience, preference), with a 4-week recall period. The OAB-SAT-q is scored by domains ranging from 0-100. Scores for the Convenience item range from 0-100. The Preference item is calculated as a percentage. Higher scores indicate higher levels of treatment satisfaction, endorsement, and convenience.

SECONDARY OUTCOMES:
Percentage of Positive Responders to Individual Treatment Satisfaction Questions 1-3 and 11 as Assessed by the OAB-SAT-q | Month 3, Month 6 and Month 12
Mean Scores on the Side Effects, Endorsement, Convenience, and Preference Domains as Assessed by the OAB-SAT-q | Month 3, Month 6 and Month 12
Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Up to Month 12
Mean Duration of Vibegron Treatment | Month 3, Month 6 and Month 12
Number of Participants Discontinuing Vibegron Treatment for the Indicated Reasons | Month 3, Month 6 and Month 12
Percentage of Participants Discontinuing Vibegron Treatment for the Indicated Reasons | Month 3, Month 6 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Urovant Sciences
Locations (64):
- United States (64):
  - Urology Centers of Alabama, Homewood, Alabama
  - 43rd Medical Associates, Phoenix, Arizona
  - Fiel Family and Sports Medicine, PC, Tempe, Arizona
  - Arkansas Urology Associates, PA, Little Rock, Arkansas
  - Golden Gate Urology, Berkley, California
  - Urology Associates of Norwalk, Norwalk, Connecticut
  - Urological Research Network, Hialeah, Florida
  - University of Florida Health Jacksonville Facility Clinic, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - South Florida Research Phase I-IV, Inc., Miami Springs, Florida
  - Tampa Urology Partners LLP, Tampa, Florida
  - Florida Urology Partners, Tampa, Florida
  - Clinical Research of Central Florida - Winter Haven, Winter Haven, Florida
  - Georgia Urology, Cartersville, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Idaho Urologic Institute, Meridian, Idaho
  - Loyola University Medical Center, Maywood, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - American Health Network of Indiana, LLC, Avon, Indiana
  - The University of Kansas Health System, Kansas City, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Owings Mills, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Valley OB-GYN Clinic, PC, Saginaw, Michigan
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - Adult & Pediatric Urology, Sartell, Minnesota
  - SVG Clinical, Las Vegas, Nevada
  - New Jersey Urology Cancer Treatment Center, Bloomfield, New Jersey
  - Lawrence OB-GYN Associates, P.C., Lawrenceville, New Jersey
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Circuit Clinical, Buffalo, New York
  - AccuMed Research Associates, Inc., Garden City, New York
  - Manhattan Medical Research Practice, PLLC, New York, New York
  - NYU Grossman School of Medicine, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - AMP Urology, Syracuse, New York
  - Atrium Health Infectious Diseases Kenilworth, Charlotte, North Carolina
  - Alliance Urology Specialists, Greensboro, North Carolina
  - FirstHealth Urogynecology, Hamlet, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Ardmore Family Practice, PA, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Obstetrics and Gynecology Associates, Inc., Cincinnati, Ohio
  - TriHealth, Cincinnati, Ohio
  - University of Cincinnati Physicians Obstetrics & Gynecology, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Institute for Female Pelvic Medicine, Allentown, Pennsylvania
  - Center for Urogynecology and Pelvic Health, King of Prussia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Southern Urogynecology, West Columbia, South Carolina
  - Urology Partners, Arlington, Texas
  - Medicus Alliance Clinical Research Organization Inc., Cedar Park, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - North Austin Urology, Round Rock, Texas
  - Medicus Alliance Clinical Research Organization Inc., Sugar Land, Texas
  - Advanced Research Institute, Ogden, Utah
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Urovant is committed to sharing participant-level data and supporting clinical documents from eligible studies with qualified external researchers. Data requests will be reviewed and approved on the basis of scientific merit. All data provided will be anonymized according to applicable laws and regulations.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be made available within 24 months after study completion and will be accessible for a time frame appropriate for the approved proposal.
Access Criteria: Access to these clinical trial data can be requested by emailing medinfo@urovant.com and will be provided following Urovant review and approval of a research proposal and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Dmochowski RR, Rovner ES, Kennelly MJ, Newman DK, Xavier K, Thomas E, Snyder D, Abedinzadeh L. Satisfaction and persistence with vibegron in the first 6 months of overactive bladder treatment: interim results of the phase 4, real-world COMPOSUR study. BMC Urol. 2025 Apr 2;25(1):66. doi: 10.1186/s12894-025-01742-6. PMID 40176006
- [Derived] Dmochowski RR, Rovner ES, Kennelly MJ, Newman DK, Abedinzadeh L, Snyder D, Thomas E, Haag-Molkenteller C, Rosenberg MT. Study design of a phase 4, real-world study (COMPOSUR) to evaluate vibegron in patients with overactive bladder. BMC Urol. 2023 Apr 24;23(1):64. doi: 10.1186/s12894-023-01240-7. PMID 37095473